CLINICAL TRIAL: NCT06805721
Title: OUTCOME in NEURORADIOLOGIA INTERVENTISTICA INDICAZIONI COMPLICANZE (ONIRIC)
Brief Title: This Three-year Observational Study Involves Patients of All Ages Undergoing Endovascular Treatment for Various Cerebral or Spinal Vascular Conditions. It Aims to Assess Pre- and Post-operative Clinical Conditions, Report Complications, and Identify Preoperative Indicators of Treatment Outcomes. Pat
Acronym: ONIRIC
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: ONIRIC
Record Dates: First submitted 2025-01-16; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Aneurysm Cerebral; AVM; DAFV; ESDC
Keywords: Endovascular treatment; Neurospychological assessment; Aneurysm; AVM; Psychological Outcome
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This three-year observational study involves patients of all ages undergoing endovascular treatment for various cerebral or spinal vascular conditions. It aims to assess pre- and post-operative clinical conditions, report complications, and identify preoperative indicators of treatment outcomes. Patients will also receive psychological support and Neuropsychological assessment. Clinical, medical, and demographic data will be recorded in a database during hospitalization and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes and any age, who are referred to the Department of Neurosurgery and Clinical Neurosciences and are candidates for interventional endovascular procedures for any cerebral or spinal pathology, will be included in the study.

Exclusion Criteria:

* /

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients of both sexes and any age who will undergo endovascular treatment and who have signed the specific consent form for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy of the Endovascular procedures | 1 year after treatment
  Describe the safety and efficacy of endovascular procedures performed for cerebro-spinal vascular diseases or hypervascularized lesions treated in the institute either through endovascular means or direct puncture. In order to the describe safety and efficay, the analysis will report the number and the nature of clinical and technical adverse events related or unrelated to a device deficiency, as assessed by CTCAE v4.0. Moreover ther will be a qualitative and quantitive (Landriel-Ibanez scale) report of the complications, and the clinical outcomes (NIHSS, mRS, Aminoff-Loug scale).
Landriel-Ibanez Scale | 1 year after treatment
  Assesses functional outcome and recovery in patients, often after neurological injuries or interventions. Scores range from 0 to 4: 0 indicates no deficits, while higher scores indicate worse functional outcomes or greater levels of disability.
National Institutes of Health Stroke Scale (NIHSS) | 1 year after treatment
  Quantifies the severity of neurological impairment in stroke patients, focusing on motor, sensory, language, and visual deficits. Scores range from 0 to 42: 0 indicates no neurological deficits, Scores 1-4 Minor stroke, Scores 5-15 Moderate stroke, Scores 16-20 Moderate-to-severe stroke, Scores 21-42 Severe stroke. Higher scores indicate greater stroke severity.
Modified Rankin Scale (mRS) | 1 year after treatment
  Assesses the degree of disability or dependence in daily activities after a stroke or other neurological conditions. Scores range from 0 to 6, with higher scores indicate worse outcomes or greater levels of disability.
Aminoff-Loug Scale | 1 year after treatment
  Evaluates functional impairments. It focuses on mobility and dependency in activities of daily living. Scores range from 0 to 5 with higher scores reflecting increasing disability and dependence in daily living activities.
Neursopychological status and Quality of life: | 1 year after treatment
  Describe the neuropsychological status and quality of life of the patient before and after (3month/6month Follow-Up and 1 year Follow-Up) the execution of such procedures. The goal is to better understand if there will be a significative change regarding such variables. The questionnaire and tests used for such assessment are listed below.
World Health Organization Disability Assessment Schedule (WHODAS): | 1 year after treatment
  Assesses disability and impairment in various life domains, with score ranging fro 0 to 100, where higher scores indicate higher disability. This scale will be part of the quality of life assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
EQ-5D-5L | 1 year after treatment
  Assesses health-related quality of life across five domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each domain has a score range fro 1 to five, where higher scores reflect lower quality of life. The VAS (Visual Analogue Scale) can be used as a quantitative measure of health outcome that reflects the patient's own judgement, with a score range from 0 ("The worst health you can imagine") to 100 ("The best health you can imagine"). This scale will be part of the quality of life assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
State and Traits Anxiety Inventory (STAI) | 1 year after treatment
  Assesses anxiety in two dimensions: state anxiety (temporary and situation-specific) and trait anxiety (a stable characteristic). Each dimension ranges from 20 to 80, with Higher scores indicate higher levels of anxiety. This scale will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Beck Depression Inventory (BDI-II) | 1 year after treatment
  Evaluates the severity of depressive symptoms. Score ranges from 0 to 63, higher scores indicate more severe depression. This scale will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Coping Orientation to Problems Experienced Inventory (Brief-COPE) | 1 year after treatment
  Evaluates coping strategies in response to stress. Each subscale ranges from 2 to 8, with different strategies assessed (e.g., active coping, avoidance), Scores indicate the extent to which specific coping strategies are used, with no direct "better" or "worse. This scale will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Mini Mental State Examination (MMSE) | 1 year after treatment
  Assessing generic cognitive function. Raw scores range from 0 to 30, according to Maesso 1993 and Magni 1996, with higher scores indicating better cognitive fuctioning. The raw score are corrected by age and educationT This test will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Raven Progressive Matrices (RPM) | 1 year after treatment
  Assees Nonverbal reasoning and problem-solving abilities. Raw Scores, according to the version of Carlesimo et. Al. 1995, range from 0 to 36, then corrected by eduction and age and converted toequivalent scores. Higher scores means better perfomance. This test will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Ray Auditory Verbal Learning Test (RAVLT) | 1 year after treatment
  Assesses verbal learning and memory. Higher scores indicate better memory performance, with lerning scores range fro 0 to 75 and log term memory from 0 to 15. Raw scores, according to the version of Carlesimo et. Al. 1996, are then corrected by age and education and converted into equivalent scores. This test will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Rey-Osterrieth Complex Figure (ROCF) | 1 year after treatment
  Assesses visuospatial ability, memory, and planning through figure reproduction and recall. Raw scores range from 0 to 36 for both reproduction and recall and, according to the version of Caffarra et. Al. 2002, are then corrected by education and age and converted to equivalent scores. Higher scores indicate better visuospatial and memory performance. This test will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Trail Making Test - A and B (TMT-A-B) | 1 year after treatment
  Measures visual attention, task-switching, and processing speed (TMT-A: sequencing numbers; TMT-B: alternating between numbers and letters). The score is determined by the time used to complete the tasks, the higher it is the poorer is the performance. Raw time scores are then corrected by age and education and then converted into equivalent scores, according to the version of Giovagnoli et al.1996. This test will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
F-A-S Phonemic Verbal Fluency Test | 1 year after treatment
  Assesses verbal fluency by generating words starting with specific letters (e.g., F, A, S) within 60 seconds. The higher is the number of words produced, the higher the performance. The raw score is then corrected by age and education and then converted into equivalent scores, according to the version of Carlesimo et al. 1995. This test will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Category Verbal Fluency Test | 1 year after treatment
  Assesses semantic verbal fluency by generating words within specific categories (e.g., animals) in 60 seconds. The higher is the number of words produced, the higher the performance. The raw score, the number of words produced in the set time, is then corrected by age and education and then converted into equivalent scores, according to the version of Carlesimo et al. 1995. This test will be part of the Neuropsychological assessment at each time point (pre intervention, post intevention, 3month Follow up, and 1 year follow up).
Verbal Digit Span | 1 year after treatment
  Assesses short term memoty (forward) and workin memory (backward). The score is determined by the amount of numers that the patiente reports correctly (span). The raw score is then corrected by age and education and then converted into equivalent scores, according to the version of Monaco et al. 2012.
Frontal Assessment Battery (FAB) | 1 year after treatment
  Assesses various executive function (Conceptualization, Mental flexibility, Motor programming, Sensitivity to interference, Inhibitory control and environmental autonomy). For each dimension the score range is from 0 to 3, resulting in a total score of 18. The raw score is then corrected by age and education and then converted into equivalent scores, according to the version of Apollnio et al. 2005.
Stroop Test | 1 year after treatment
  The test consist of three different parts (words, color and word-color) and assesses processing speed, attention and inhibitory control. The performance is determined by time and errrors in completing the task. Both time and errors raw scores, after being processed through the dedicated formula, are then corrected by age and education and the converted in equivalent scores, according to Cafarra et al. 2002.

SECONDARY OUTCOMES:
Preprocedural outcome identification | pre-procedure
  Identify the pre-procedural indicators of outcome in the various treated pathologies. The analysis will include a report of the possible association between the pre procedural indicators (socio-demographic variables, comorbidities, pre-procedure medical treatment, morphology, dimension and location of the endovascular pathology) and the clinical and neuropsychological outcome describe above.
Socio-demographic variables | pre-procedure
  Age in years, Sex, education in years
Comorbidities | pre-procedure
  Hypertension, smoker, diabete, familiarity with endovascular pathololgies.
Pre-procedure medical treatment | pre-procedure
  It will be reported if the patient will be in single antiplatelet or dual antiplatelet medication before the procedure and the wich drug is used.
Morphology of the endovascular pathology | pre-procedure
  In case of aneurysm, it will report the if the morphology is saccular, dissecant, ovalar, fusiform, with a large or a small collar.
  In case of MAV, the morphology will be described using the Spetzler-Martin scale(0-5 points): size (0-3 points, venous drainage (0-1 point), eloquent brain areas (0-1 point), grading (0-1 Point).
Dimension in mm | pre-procedure
  It will report the dimension of the pathology (AVMS, SDH, Aneurysm, FAVD, FAVDs)
Location | pre-procedure
  The location will include the hemisphere side (left, right, bilateral) and the information about witch artery/vein is involved in the pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Carlo Besta Neurological Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No